CLINICAL TRIAL: NCT06719635
Title: Laparoscopic Presacral Neurectomy Versus Fluoroscopically Guided Superior Hypogastric Plexus Neurolysis for Treatment of Chronic Pelvic Pain: A Double-Blind, Randomized Controlled Trial.
Brief Title: Management Modalities of Chronic Pelvic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pelvic Pain Management
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Presacral Neurectomy (Active Comparator): The patients will undergo Laparoscopic Presacral Neurectomy under general anesthesia.
  Interventions: Procedure: Laparoscopic Presacral Neurectomy
- Fluoroscopically guided Superior Hypogastric Neurolysis (Active Comparator): The patients will receive fluoroscopically guided Superior Hypogastric Plexus Neurolysis with Radiofrequency of the Sacral Roots 2,3,4.
  Interventions: Procedure: Fluoroscopically guided Superior Hypogastric Plexus Neurolysis

INTERVENTIONS:
Procedure: Laparoscopic Presacral Neurectomy — Laparoscopy will be performed under general anesthesia. Then, nerve plexuses will be identified and freed from their underlying tissue, which contains the left common iliac and middle sacral veins. This will be followed by cauterization and cutting of the nerve plexuses.
  Arms: Laparoscopic Presacral Neurectomy
Procedure: Fluoroscopically guided Superior Hypogastric Plexus Neurolysis — The patients will receive fluoroscopically guided Superior Hypogastric Plexus Neurolysis using 3 mL of 75% ethanol and Radiofrequency of the Sacral nerve Roots 2-4.
  Arms: Fluoroscopically guided Superior Hypogastric Neurolysis

SUMMARY:
Chronic pelvic pain remains a challenging disorder to treat because of the complexities of pain sensation and unclear etiology. Standard medical and surgical treatments seldom prove effective at improving quality of life and pain intensity among affected women.

DETAILED DESCRIPTION:
Chronic pelvic pain remains a challenging disorder to treat because of the complexities of pain sensation and unclear etiology. Standard medical and surgical treatments seldom prove effective at improving quality of life and pain intensity among affected women. The current study will investigate whether Laparoscopic Presacral Neurectomy or Fluoroscopically Guided Superior Hypogastric Plexus Neurolysis is more effective for treating chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Body mass index < 35 kg/m2.
* Adult patients with chronic pelvic and perineal pain due to pelvic cancer.
* Visual Analog Scale pain score ≥ 5 on a 0-10 scale despite treatment with a standard analgesic.

Exclusion Criteria:

* Uncooperative patient.
* Patients with coagulopathy, infection at the site of injection, severe cardiac compromise, or intolerance to sympathetic block.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-12-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain score | At the end of the first month after the procedure.
  The percentage of patients who achieved > 50% decline in their Visual analogue pain score "from the baseline value" before intervention at the end of the first month.

SECONDARY OUTCOMES:
Daily analgesic requirements | At the end of the first 2 weeks, 1st month, 2nd month, 3rd month, and 6th month after the procedure.
  Daily analgesic requirements at the end of the first 2 weeks, 1st month, 2nd month, 3rd month, and 6th month after the procedure.
Associated adverse events | At the end of the first month after the procedure.
  Any related adverse events "e.g. hypotension, bleeding or neurological deficits" in the first month after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Abdalla Mohamed Gouda, MD, Principal Investigator — Department of Anesthesia, Intensive Care & Pain Management, Zagazig University
Locations (1):
- Zagazig university hospital, Zagazig, Al-Sharkia, Egypt

REFERENCES:
- [Background] de Leon-Casasola OA, Kent E, Lema MJ. Neurolytic superior hypogastric plexus block for chronic pelvic pain associated with cancer. Pain. 1993 Aug;54(2):145-151. doi: 10.1016/0304-3959(93)90202-Z. PMID 8233527
- [Background] Ghai V, Subramanian V, Jan H, Pergialiotis V, Thakar R, Doumouchtsis SK; CHORUS: An International Collaboration for Harmonising Outcomes, Research, Standards in Urogynaecology, Women's Health. A systematic review on reported outcomes and outcome measures in female idiopathic chronic pelvic pain for the development of a core outcome set. BJOG. 2021 Mar;128(4):628-634. doi: 10.1111/1471-0528.16412. Epub 2020 Sep 1. PMID 32654406
- [Background] Hetta DF, Mohamed AA, Abdel Eman RM, Abd El Aal FA, Helal ME. Pulsed Radiofrequency of the Sacral Roots Improves the Success Rate of Superior Hypogastric Plexus Neurolysis in Controlling Pelvic and Perineal Cancer Pain. Pain Physician. 2020 Mar;23(2):149-157. PMID 32214294
- [Background] Soysal ME, Soysal S, Gurses E, Ozer S. Laparoscopic presacral neurolysis for endometriosis-related pelvic pain. Hum Reprod. 2003 Mar;18(3):588-92. doi: 10.1093/humrep/deg127. PMID 12615830